CLINICAL TRIAL: NCT02590341
Title: Myocarditis Registry for Children and Adolescents - MYKKE
Acronym: MYKKE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Collaborators: Competence Network for Congenital Heart Defects (Other Government)
Responsible Party: Sponsor
Other Study IDs: MYKKE Registry
Record Dates: First submitted 2015-10-08; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Myocarditis
Keywords: myocarditis; children; adolescents; registry; multi-center; pediatric; heart failure; inflammatory heart disease; inflammatory cardiomyopathy
MeSH Terms: conditions — Myocarditis; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
MYKKE is a prospective multi-center registry for children and adolescents with myocarditis. The aim is to generate prospective multi-center data on epidemiology, diagnostics, and therapy of pediatric patients with myocarditis in order to enable evidence-based diagnostic and therapeutic approaches for this myocardial disease.

DETAILED DESCRIPTION:
MYKKE is a long-term prospective registry providing a core platform for clinical research studies, which can be attached in a modular fashion. After a six-month pilot phase including 8 centers, the basic registry was opened in June 2014 to all hospitals in Germany treating patients with paediatric heart disease. While the scientific lead is with two study coordinators and a study group consisting of principal investigators from the collaborating centres ("MYKKE Investigators"), MYKKE is hosted and technically administered by the Competence Network for Congenital Heart Defects, which was initiated in 2003 by the Federal Ministry of Education and Research of the German government and is now part of the German Center for Cardiovascular Research (DZHK). Ethical approval was first obtained at the initiating centre (Deutsches Herzzentrum Berlin) and subsequently confirmed by local authorities of all collaborating centres.

The treating physicians enter basic data from patients enrolled at the study site via an online web interface to a central study database. For each patient, a specific patient identification number (PID) is generated based on name, first name and date of birth in order to store data in a pseudonymized fashion. As the PIDs are generated by a specific algorithm, data from the same patient are always linked to the same dataset even when data from different visits are entered by different institutions.

The web interface provides two different forms for each patient. The first form ("general sheet") is filled-in only at first presentation and consists of 12 items regarding disease and patient history, and initial symptoms of the disease. The second type of sheet ("current visit") can be generated once for each new patient visit and includes 52 items on characteristics of the current visit, current symptoms, diagnostic tests performed, confidence of the treating physician in the diagnosis on a subjective scale, left-ventricular function, therapy, complications, and follow-up care provider after discharge. Items primarily require yes/no responses via ticking respective boxes, allowing for completing each data sheet in <5 minutes when all data are available.

ELIGIBILITY:
Inclusion Criteria:

* Admission or referral diagnosis of myocarditis
* Age <18 years
* Written informed consent of the parents or legal guardians

Exclusion Criteria:

* Unwillingness to give consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients admitted to pediatric heart centers or pediatric cardiology departments
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-06; Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year
admission for heart failure | one year
major cardiovascular events | one year
  cardiovascular death, need for mechanical ventricular support or heart transplantation, sustained ventricular arrhythmia, decompensated heart failure requiring catecholamine therapy

SECONDARY OUTCOMES:
systolic dysfunction | one year
  left ventricular ejection fraction <50%
diastolic dysfunction | one year
  elevated natriuretic peptides, E/E' >15, left ventricular ejection fraction >= 50%
impaired exercise tolerance | one year
  maximal oxygen uptake (VO2max) <5th percentile of normal

OTHER OUTCOMES:
medium-term all cause mortality | five years
  mortality due to all causes at 5 years
long-term all cause mortality | ten years
  mortality due to all causes at 10 years
medium-term admission for heart failure | five years
  admission for heart failure at 5 years
long-term admission for heart failure | ten years
  admission for heart failure at 10 years
medium-term major cardiovascular events | five years
  major cardiovascular events at 5 years (cardiovascular death, need for mechanical ventricular support or heart transplantation, sustained ventricular arrhythmia, decompensated heart failure requiring catecholamine therapy)
long-term major cardiovascular events | ten years
  major cardiovascular events at 10 years (cardiovascular death, need for mechanical ventricular support or heart transplantation, sustained ventricular arrhythmia, decompensated heart failure requiring catecholamine therapy)
medium-term systolic dysfunction | five years
  left ventricular ejection fraction <50%
long-term systolic dysfunction | ten years
  left ventricular ejection fraction <50%
medium-term diastolic dysfunction | five years
  elevated natriuretic peptides, E/E' >15, left ventricular ejection fraction >=50%
long-term diastolic dysfunction | ten years
  elevated natriuretic peptides, E/E' >15, left ventricular ejection fraction >=50%
medium-term impaired exercise tolerance | five years
  maximal oxygen uptake (VO2max) <5th percentile of normal
long-term impaired exercise tolerance | ten years
  maximal oxygen uptake (VO2max) <5th percentile of normal

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Messroghli, MD, Study Director — German Heart Institute; Stephan N Schubert, MD, Study Director — German Heart Institute
Locations (13):
- Germany (13):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Charite - Universitätsmedizin Berlin, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Klinikum Links der Weser, Bremen
  - Universitätsklinikum Erlangen, Erlangen
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Freiburg im Breisgau
  - Universitätsklinikum Giessen und Marburg, Giessen
  - Universitätsmedizin Göttingen, Göttingen
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Schleswig-Holstein, Kiel

REFERENCES:
- [Derived] Seidel F, Nygren TM, Opgen-Rhein B, Hecht T, Boehne M, Weickmann J, Anderheiden F, Reineker K, Bocker D, Rentzsch A, Wiegand G, Fischer M, Kiski D, Frede W, Ruf B, Tarusinov G, Papakostas K, Logeswaran T, Schiebel A, Voges I, Kaestner M, Kramp J, Kerst G, Khedim M, Gatzweiler E, Wannenmacher B, Knirsch W, Meyer-Dobkowitz L, Donner B, Klingner J, Rau C, Haller S, Brinkmann A, Nitsche A, Noldt M, Schmoock G, Herzmann C, Degenhardt U, Buhler S, Enders M, Hermes J, Rolfs N, Manuylova T, Schwarzkopf E, Beudt J, Siffczyk C, Schubert S, Sandfort M, Klingel K. Severe Myocarditis Increase in Children Associated With Parvovirus B19 Infection: MYKKE Registry and German Surveillance Data. JACC Heart Fail. 2025 Dec 29:102854. doi: 10.1016/j.jchf.2025.102854. Online ahead of print. PMID 41493405
- See also: Website of MYKKE registry (German language only) — http://mykke.de